CLINICAL TRIAL: NCT03600246
Title: Prospective Observational Registry for Obstructive Sleep Apnea in Patients With Acute Myocardial Infarction
Acronym: OSAAMI
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun-Won Lee, Assistant professor, Wonju Severance Christian Hospital
Other Study IDs: WATCHPAT-AMI
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Sleep Apnea; Acute Myocardial Infarction
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: WATCH-PAT — WatchPAT is an FDA-approved portable diagnostic device that uniquely uses finger based physiology and innovative technology to enable simple and accurate Obstructive Sleep Apnea (OSA) testing while avoiding the complexity and discomfort associated with traditional air-flow based systems.

SUMMARY:
Obstructive sleep apnea (OSA) has been known as a risk factor for coronary artery disease, heart failure, cerebrovascular accident and atrial fibrillation. One study reported that patients with OSA have more atherosclerotic plaque burden in intravascular ultrasonography examination. Among patients who admitted with acute myocardial infarction (AMI), 65.7% (69 of 105) patients were diagnosed with OSA. Other long-term follow-up study revealed that 45.4% of patients (594 of 1311) who performed percutaneous coronary intervention (PCI) were diagnosed with OSA. Moreover, the OSA group was a significant independent predictor of major adverse cardiac and cerebrovascular events (MACCEs).

Polysomnography (PSG) is the gold standard for the diagnosis of OSA. But, PSG is expensive, time-consuming and difficult to perform immediately. Recently, a portable device named WATCH-PAT (Itamar Ltd, Israel) was developed for the diagnosis of OSA. Validation study demonstrated a high correlation between WATCH-PAT and PSG in apnea-hypopnea index, lowest oxygen saturation and sleep time. This result suggested WATCH-PAT can be performed as an alternative or supportive device of PSG. WATCH-PAT. The portable device also can be useful to detect OSA in bus drivers who can be the reason for public traffic accidents. Moreover, WATCH-PAT can be applied to assess postoperative improvement of OSA.

Although OSA is known as one of the risk factors for cardiovascular disease, there is a lack of evidence to recommend of the evaluation of sleep disorder in patient with coronary artery disease. Awareness and compliance for OSA are very low in both patients and cardiologists. Active diagnosis and treatment are definitely needed. Therefore, the primary endpoint of this study is to evaluate the prevalence of OSA in AMI patients who treated PCI. The secondary endpoint is to evaluate the 1-year incidence rate of MACCEs according to the presence or absence of OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 years
2. Successful PCI in at least one major epicedial coronary artery

Exclusion Criteria:

1. IABP or other hemodynamic support device
2. Known OSA on CPAP treatment
3. Intubation for mechanical ventilation
4. Sedation given before WATCH-PAT study
5. Cardiogenic shock (SBP<90mmHg)
6. Heart failure requiring oxygen supplement
7. High risk of malignant ventricular arrhythmia
8. Pregnancy
9. History of malignancy
10. Expected life span <12 months
11. Inability to provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with acute myocardial infarction and treated percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA (%) | 1 day during sleep
  Incidence rate (%) of obstructive sleep apnea

SECONDARY OUTCOMES:
MACCE (%) | 1 year
  Incidence rate (%) of MACCE defined as composite endpoint of all-cause death, myocardial infarction, any revacularization and stroke
All-cause death (%) | 1 year
  Incidence rate (%) of all-cause death
Any myocardial infarction (%) | 1 year
  Incidence rate (%) of any myocardial infarction
Any revascularization (%) | 1 year
  Incidence rate (%) of any revascularization
Stroke (%) | 1 year
  Incidence rate (%) of stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Won Lee, MD, Principal Investigator — Assistant professor
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, South Korea

IPD SHARING:
Plan to Share IPD: No